CLINICAL TRIAL: NCT00618995
Title: A Randomized, Double-Blind, Placebo-Controlled, 4-Period, Crossover Study to Evaluate the Effects of ER Niacin/Laropiprant, Laropiprant, ER Niacin, and Placebo on Urinary Prostanoid Metabolites in Subjects With Type 2 Diabetes
Brief Title: A Study to Evaluate the Effects of ER Niacin/Laropiprant, Laropiprant, ER Niacin, and Placebo on Urinary Prostanoid Metabolites (0524A-079)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-079; 2008_508
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Results first posted 2009-02-05 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- A (Experimental): Arm A: ER niacin/laropiprant + Placebo to laropiprant
  Interventions: Drug: Comparator: ER niacin (+) laropiprant
- B (Experimental): Arm B: ER niacin + Placebo to laropiprant
  Interventions: Drug: Comparator: ER niacin
- C (Experimental): Arm C: laropiprant + Placebo to ER Niacin/laropiprant
  Interventions: Drug: Comparator: laropiprant
- D (Placebo Comparator): Arm D: Placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: Comparator: ER niacin (+) laropiprant — ER niacin 2 g/ laropiprant 40 mg daily for 7 days.
  Arms: A
Drug: Comparator: ER niacin — ER niacin 2 g daily for 7 days.
  Arms: B
Drug: Comparator: laropiprant — laropiprant 40 mg daily for 7 days.
  Arms: C
Drug: Comparator: placebo — matching placebo tablets for each of the interventions once daily for 7 days
  Arms: D

SUMMARY:
The purpose of this study is to evaluate the potential effects of ER niacin/laropiprant, ER niacin, laropiprant, and placebo over the course of seven days on urinary levels of a specific metabolite (which is a marker of in vivo platelet reactivity).

DETAILED DESCRIPTION:
Subjects will receive 1 of 4 treatments per period and will eventually receive all 4 treatments:

Treatment A: ER niacin 2g/laropiprant 40 mg daily + Placebo to laropiprant for 7 days

Treatment B: ER niacin 2 g daily + Placebo to laropiprant for 7

days

Treatment C: laropiprant 40 mg daily + Placebo to ER niacin/laropiprant for 7 days

Treatment D: placebo daily for 7 days. There will be at least a 7-day interval between dosing on Day 7 of a period and dosing on Day 1 of the subsequent period

ELIGIBILITY:
Inclusion Criteria:

* Female subjects may not be pregnant and/or will agree to use appropriate method of contraception beginning at least 2 weeks prior to administration of the first dose of study drug in the first treatment period, throughout the study and until at least 2 weeks after administration of the last dose of study drug in the last treatment period
* Subject has a history of T2DM either treated with diet and exercise alone or with metformin or a sulfonylurea
* Subject is judged to be in good health (other than history of Type 2 diabetes mellitus) based on medical history, physical examination, vital sign measurements, and laboratory safety tests performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug
* Subject has no clinically significant abnormality on electrocardiogram (ECG) performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug
* Subject has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months; subjects who have discontinued smoking or the use of nicotine/nicotine containing products for at least approximately 3 months may be enrolled in the study at the discretion of the investigator

Exclusion Criteria:

* Subject is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder over the last 5 to 10 years
* Subject has a history of stroke, chronic seizures, or major neurological disorder
* Subject has a history of clinically significant endocrine (except for Type 2 diabetes mellitus), gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Subject has a history of neoplastic disease (including leukemia, lymphoma, malignant melanoma), or myeloproliferative disease, regardless of the time since treatment
* Subject has history of a blood or platelet related disorder including prior deep venous thrombosis. Subject is being treated with coumadin, heparin, clopidogrel or has used these agents within 2 weeks of screening. Subject is being treated with aspirin or has used this agent within 3 weeks prior to administration of screening
* Subject is unable to refrain from or anticipates the use of any medication (with the exception of metformin or sulfonylurea agents), including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks until the post-study visit. No concomitant medications may be taken during the study
* Subject consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages, per day
* Subject consumes excessive amounts, defined as greater than 6, of coffee, tea, cola, or other caffeinated beverages per day
* Subject has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks prior to the prestudy (screening) visit
* Subject has a history of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Subject uses insulin, PPAR gamma agonists (rosiglitazone or pioglitazone), exenatide (Byetta), acarbose (Prandase, Precose) or dipeptidyl-peptidase 4 (DPP-4) inhibitors (JANUVIA™1)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lauring B, Dishy V, Luo WL, Laterza O, Patterson J, Cote J, Chao A, Larson P, Gutierrez M, Wagner JA, Lai E. Laropiprant in combination with extended-release niacin does not alter urine 11-dehydrothromboxane B2, a marker of in vivo platelet function, in healthy, hypercholesterolemic, and diabetic subjects. J Clin Pharmacol. 2009 Dec;49(12):1426-35. doi: 10.1177/0091270009339593. Epub 2009 Oct 15. PMID 19833861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I
  First Patient Enrolled 21 Aug 2007, First Patient Treated 7 Sept 2007.
  Study conducted at 3 centers: Arkansas Research Medical Testing, LLC, Little Rock, AR; Healthcare Discoveries Inc., San Antonio, TX; and Comprehensive Phase One, Fort Myers, FL. Merck's ER Niacin was used.
Pre-assignment Details: Subjects were treated either w/diet and exercise alone, or with metformin, or a sulfonylurea, and had to be on stable meds for >= 8 wks pre-study.
Groups:
- Sequence 1: D/C/A/B; Sequence 2: C/B/D/A; Sequence 3: B/A/C/D; Sequence 4: A/D/B/C: A = ER Niacin 2 g/Laropiprant 40 mg once daily for 7 days
  B = ER Niacin 2 g once daily for 7 days
  C = Laropiprant 40 mg once daily for 7 days
  D = Placebo once daily for 7 days
Period: Period 1
Arm/Group | Sequence 1: D/C/A/B | Sequence 2: C/B/D/A | Sequence 3: B/A/C/D | Sequence 4: A/D/B/C
Started | 6 | 7 | 7 | 6
Completed | 6 | 6 | 5 | 6
Not Completed | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Period: Period 2
Arm/Group | Sequence 1: D/C/A/B | Sequence 2: C/B/D/A | Sequence 3: B/A/C/D | Sequence 4: A/D/B/C
Started | 6 | 6 | 5 | 6
Completed | 6 | 6 | 4 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Period: Period 3
Arm/Group | Sequence 1: D/C/A/B | Sequence 2: C/B/D/A | Sequence 3: B/A/C/D | Sequence 4: A/D/B/C
Started | 6 | 6 | 4 | 6
Completed | 6 | 6 | 4 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1: D/C/A/B | Sequence 2: C/B/D/A | Sequence 3: B/A/C/D | Sequence 4: A/D/B/C
Started | 6 | 6 | 4 | 6
Completed | 5 | 6 | 4 | 6
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Totals For Study: All participants in the study.
Arm/Group | Totals For Study
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Height [Mean (Full Range); unit: cm] | 163.9 [150 to 181.5]
Weight [Mean (Full Range); unit: kg] | 85.9 [55.0 to 127.2]
urinary 11-dTxB2 [Median (Full Range); unit: pg/mg creatinine] — urinary levels of 11-dehydrothromboxane B2 (24-hour collection)
  pg/mg creatinine | 639.1 [304.5 to 1045.6]
urinary PGI2-Metabolite [Median (Full Range); unit: pg/mg creatinine] — urinary levels of 2,3-dinor 6-keto-PGF1a (Prostaglandin I-M) 24 hour collection
  pg/mg creatinine | 167.5 [79.4 to 356.0]

OUTCOME MEASURES:

1. Primary Outcome: Urinary 11-Dehydrothromboxane B2 (11-dTxB2)
Description: The creatinine-normalized urine levels of 11-dTxB2 on Day 7 following a 7 day course of daily dosing in the overall 24 hour collection interval
Time Frame: On Day 7 across the 24-hour urinary collection period.
Population: Twenty-six (26) subjects (including replacements) were enrolled in this study. All available subjects (besides the 2 that were excluded due to suspected NSAID/Aspirin use) who complied with the protocol and had partial data were included in the subsequent statistical analysis models/comparisons.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg creatinine
Groups:
- ER Niacin/Laropiprant: Extended Release (ER) Niacin 2 g/Laropiprant 40 mg once daily for 7 days
- ER Niacin: ER Niacin 2 g once daily for 7 days
- Laropiprant: Laropiprant 40 mg once daily for 7 days
- Placebo: Placebo once daily for 7 days
Arm/Group | ER Niacin/Laropiprant | ER Niacin | Laropiprant | Placebo
Number analyzed (Participants) | 22 | 21 | 22 | 22
pg/mg creatinine | 525.3 [423.8 to 651.1] | 540.8 [435.0 to 672.3] | 585.3 [472.2 to 725.4] | 625.1 [504.3 to 774.8]
Statistical Analysis 1: Comparison: ER Niacin/Laropiprant vs ER Niacin; The endpoint is the urine levels of 11-dTxB2 on Day 7 following a 7 day course of daily dosing in the overall 24 hour collection interval. The point estimate and 90% confidence intervals (CIs) were calculated for the geometric mean ratio (GMR) [Treatment A/B] of the urine levels of 11-dTxB2 on Day 7; Test type: Non-Inferiority or Equivalence — Two treatments are comparable if the geometric mean ratio (GMR) is contained within the interval [0.50-2.00]; Geometric least-squares mean ratio = 0.97, 90% CI [0.8 to 1.18]
Statistical Analysis 2: Comparison: Laropiprant vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.94, 90% CI [0.77 to 1.14]
Statistical Analysis 3: Comparison: ER Niacin vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.87, 90% CI [0.71 to 1.05]
Statistical Analysis 4: Comparison: ER Niacin/Laropiprant vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.84, 90% CI [0.69 to 1.02]
Statistical Analysis 5: Comparison: ER Niacin vs Laropiprant; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.92, 90% CI [0.76 to 1.13]
Statistical Analysis 6: Comparison: ER Niacin/Laropiprant vs Laropiprant; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.9, 90% CI [0.74 to 1.09]

2. Secondary Outcome: Prostaglandin I Metabolite (PGI-M)
Description: PGI-M in the Overall 24 Hour Collection Interval Following Administration on Day 7
Time Frame: On Day 7 across the 24-hour urinary collection period.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg creatinine
Arm/Group | ER Niacin/Laropiprant | ER Niacin | Laropiprant | Placebo
Number analyzed (Participants) | 22 | 21 | 22 | 22
pg/mg creatinine | 90.1 [74.5 to 109.0] | 95.4 [78.7 to 115.5] | 158.5 [131.0 to 191.8] | 168.1 [139.0 to 203.4]
Statistical Analysis 1: Comparison: ER Niacin/Laropiprant vs ER Niacin; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.94, 90% CI [0.84 to 1.06]
Statistical Analysis 2: Comparison: Laropiprant vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.94, 90% CI [0.84 to 1.05]
Statistical Analysis 3: Comparison: ER Niacin vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.57, 90% CI [0.51 to 0.64]
Statistical Analysis 4: Comparison: ER Niacin/Laropiprant vs Placebo; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.54, 90% CI [0.48 to 0.60]
Statistical Analysis 5: Comparison: ER Niacin vs Laropiprant; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.60, 90% CI [0.54 to 0.67]
Statistical Analysis 6: Comparison: ER Niacin/Laropiprant vs Laropiprant; Test type: Superiority or Other; Geometric least-squares mean ratio = 0.57, 90% CI [0.51 to 0.64]

ADVERSE EVENTS:
Arm/Group | ER Niacin/Laropiprant | ER Niacin | Laropiprant | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/25 | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 17/23 | 23/25 | 12/23 | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ER Niacin/Laropiprant (N=23) | ER Niacin (N=25) | Laropiprant (N=23) | Placebo (N=22)
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ER Niacin/Laropiprant (N=23) | ER Niacin (N=25) | Laropiprant (N=23) | Placebo (N=22)
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 3 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 1 | 2
Nausea (Gastrointestinal disorders) | 4 | 9 | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 4 | 1 | 1
Asthenia (General disorders) | 0 | 2 | 2 | 0
Feeling Hot (General disorders) | 1 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Burning Sensation (Nervous system disorders) | 2 | 6 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 1 | 0
Headache (Nervous system disorders) | 3 | 6 | 4 | 4
Paraesthesia (Nervous system disorders) | 2 | 4 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 6 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 14 | 2 | 3
Flushing (Vascular disorders) | 7 | 17 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.